CLINICAL TRIAL: NCT05566067
Title: Survey of Anesthesiology Residents' Perceptions of Critical Care Medicine as a Career at One Academic Center
Brief Title: Survey of Anesthesiology Residents' Perceptions of Critical Care Medicine as a Career
Status: Not yet recruiting | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Chi-Ho Ban Tsui, Professor-Med Ctr Line, Stanford University
Other Study IDs: 67638
Record Dates: First submitted 2022-09-29; First posted 2022-10-04 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Anesthesia
Keywords: critical care medicine; fellowship; anesthesiology residency; perception; anesthesia
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Anesthesiology residents: We plan to distribute a survey to the Stanford anesthesiology residents to investigate the factors that influence residents' decision to pursue a career as a critical care physician.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — There will be no interventions for study participants. Participants will be asked to complete a survey.

SUMMARY:
This study's goal is to investigate the reasons behind the decline in interest in critical care fellowships among anesthesia residents.

DETAILED DESCRIPTION:
Anesthesia-based critical care medicine (CCM) is at a crossroads at the turn of the millennium. Although anesthesiologists were pioneers in the field of critical care, their surgical and pulmonary medicine counterparts have now eclipsed them in terms of both numbers and influence. In the United States, anesthesia-based CCM is a niche specialization of anesthesiology, while in Europe, anesthesiologists play a central role in critical care. Anesthesia-based critical care physician production has remained low on an annual basis. Some medical students join anesthesiology residencies with an interest in critical care training, but this enthusiasm appears to diminish as the number of years of residency grows. In the United States, anesthesiology residents have been unable to fill many critical care fellowship spots consistently. This survey aims to investigate the factors that influence residents' decision to pursue a career as a critical care physician, as it is essential to comprehend the underlying reasons for such a decline.

ELIGIBILITY:
Inclusion Criteria:

* Anesthesiology residents at Stanford

Exclusion Criteria:

* Non-anesthesiology residents at Stanford

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Anesthesiology residents at Stanford
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Decline in applying to CCM fellowships | 3 months
  Examining the declining applying to CCM fellowship whether due to intrinsic factors (i.e., nature of CCM practice) vs extrinsic factors (i.e., job market and relative competing compensation)

CONTACTS AND LOCATIONS:
Overall Officials: Ban CH Tsui, MD, Study Director — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hanson CW 3rd, Durbin CG Jr, Maccioli GA, Deutschman CS, Sladen RN, Pronovost PJ, Gattinoni L. The anesthesiologist in critical care medicine: past, present, and future. Anesthesiology. 2001 Sep;95(3):781-8. doi: 10.1097/00000542-200109000-00034. No abstract available. PMID 11575554